CLINICAL TRIAL: NCT04610476
Title: A Prospective, Randomized, Controlled, Open Label, Assessor-blinded, Parallel-group Phase III Clinical Trial to Evaluate the Impact of Tapering Systemic Immunosuppressive Therapy in a Treat-to-target Approach on Maintaining Minimal Disease Activity in Adult Subjects With Psoriatic Arthritis
Brief Title: Impact of Tapering Immunosuppressants on Maintaining Minimal Disease Activity in Adult Subjects With Psoriatic Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKER-ATTRACTOR -01
Record Dates: First submitted 2020-09-18; First posted 2020-10-30 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Psoriatic Arthritis; Withdrawal; Reduction
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Prednisolone; Sulfasalazine; Leflunomide; Methotrexate; tofacitinib; apremilast; Etanercept; Adalimumab; Infliximab; Certolizumab Pegol; golimumab; Abatacept; secukinumab; ixekizumab; Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Individual previous stable glucocorticoid/DMARD therapy is continued
- Reduction group (Experimental): Individual previous stable dosage of glucocorticoids/DMARDs will be stepwise reduced according to a predefined algorithm
  Interventions: Drug: Prednisolone; Drug: Sulfasalazine; Drug: Leflunomide; Drug: Methotrexate; Drug: Tofacitinib; Drug: Apremilast; Drug: Etanercept; Drug: Adalimumab; Drug: Infliximab; Drug: Certolizumab pegol; Drug: Golimumab; Drug: Abatacept; Drug: Secukinumab; Drug: Ixekizumab; Drug: Ustekinumab

INTERVENTIONS:
Drug: Prednisolone — Prednisolone oral 1-5 mg/day
  Other Names: Prednisolone generic drugs
  Arms: Reduction group
Drug: Sulfasalazine — Sulfasalazine oral 2 x 1000 mg/day
  Other Names: Azulfidine
  Arms: Reduction group
Drug: Leflunomide — Leflunomide oral 20 mg/day
  Other Names: Arava
  Arms: Reduction group
Drug: Methotrexate — Methotrexate oral > 10 - 30 mg/ week/ 10 mg/week/ 7.5 mg/week; s.c. 15 (7.5 -25) mg/week
  Other Names: Lantarel, Metex
  Arms: Reduction group
Drug: Tofacitinib — Tofacitinib oral 2 x 5 mg/day/ 1 x 5 mg/day/11 mg/day
  Other Names: Xeljanz
  Arms: Reduction group
Drug: Apremilast — Apremilast oral 2 x 30 mg/day/1 x 30 mg/day
  Other Names: Otezla
  Arms: Reduction group
Drug: Etanercept — Etanercept s.c. 2 x 25 mg /week OR 1 x 50 mg/week
  Other Names: Enbrel, Erelzi, Benepali
  Arms: Reduction group
Drug: Adalimumab — Adalimumab s.c. 40 mg every 2 weeks
  Other Names: Humira, Amgevita, Imraldi, Hyrimoz
  Arms: Reduction group
Drug: Infliximab — Infliximab i.v. 5 mg/kg BW every 8 weeks
  Other Names: Remicade, Zessly, Inflectra
  Arms: Reduction group
Drug: Certolizumab pegol — Certolizumab pegol s.c. 1x 200 mg every 2 weeks/1x400 mg every 4 weeks
  Other Names: Cimzia
  Arms: Reduction group
Drug: Golimumab — Golimumab s.c. 1x 50 mg every 4 weeks
  Other Names: Simponi
  Arms: Reduction group
Drug: Abatacept — Abatacept s.c. 1x125 mg/week OR Abatacept i.v. 500-1000mg (adapted to BW) every 4 weeks
  Other Names: Orencia
  Arms: Reduction group
Drug: Secukinumab — Secukinumab s.c.1x 150 mg OR 1x 300 mg every 4 weeks
  Other Names: Cosentyx
  Arms: Reduction group
Drug: Ixekizumab — Ixekizumab s.c. 1x 80 mg every 4 weeks
  Other Names: Taltz
  Arms: Reduction group
Drug: Ustekinumab — Ustekinumab s.c. Maintenance dose 1x45 mg every 12 weeks
  Other Names: Stelara
  Arms: Reduction group

SUMMARY:
The rationale for this study is to investigate whether in psoriatic arthritis (PsA) patients in stable remission a reduction or complete discontinuation of immunosuppressive therapy can be achieved in a treat-to-target approach while maintaining in remission. Due to the lack of reliable data that answers the question of how to safely reduce medication in which patients, this study will test a pragmatic treatment algorithm that can be applied in clinical practice and that offers a gradual reduction with escape strategies in order to facilitate the maintenance of remission.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject
* Understanding of study procedures and willingness to abide by all procedures during the course of the study.
* Adult subject; age range 18-≤75 years
* Male or female subject
* Diagnosis of PsA according to CASPAR criteria
* Disease status "MDA" for at least 6 months
* Subject should have been treated without alterations of therapy (fixed dose and drug) for at least 6 months with one or more of the following drugs:

  i. csDMARD Leflunomid (e.g. Arava), Sulfasalazin (e.g. Azulfidine RA, Pleon RA), Methotrexate (e.g. Lantarel, Metex) AND/OR ii. bDMARD/tsDMARD: Etanercept (e.g. Enbrel, Erelzi, Benepali), Adalimumab (e.g. Humira, Amgevita, Imraldi, Hyrimoz), Infliximab (e.g. Remicade, Zessly, Inflectra), Golimumab (Simponi), Certolizumab (Cimzia), Abatacept (Orencia), Apremilast (Otezla), Ustekinumab (Stelara), Secukinumab (Cosentyx), Ixekizumab (Taltz), Tofacitinib (Xeljanz) AND/OR (c) glucocorticoids (≤5mg prednisolone equivalent).
* Women of childbearing potential must be using a highly effective method of birth control.
* Male subjects using an adequate contraceptive method at the investigator's discretion.

Exclusion Criteria:

* Diagnosis of any other rheumatological/ immunological disease such as rheumatoid arthritis, SLE, PSS, MCTD, M. Behcet or M. Wegener
* Concomitant florid (not sufficiently adjusted under treatment) autoimmune disease such as autoimmune hepatitis or Hashimoto's disease
* Use of any inadmissible medication (e.g. current treatment with DMARDs other than mentioned above or drugs under development)
* Treatment with systemic glucocorticoids (daily dose >5mg prednisolone equivalent) during the last 6 months before randomization. Intra-articular or entheseal injections of glucocorticoids do not constitute an exclusion criterion
* Malignant disease currently under oncological treatment or history of a recent malignancy with moderate or high risk of relapse within 5 years prior to Screening
* Existence of another disease including the presence of laboratory abnormalities which, at the discretion of the investigator, would result in a disproportionate risk to the patient concerned or confounds the ability to interpret data from the study
* Any anti-inflammatory (excluding NSAIDs) or immunosuppressive therapy for other reasons than PsA or psoriasis during the last 3 months before Screening
* Nursing mother or pregnant woman as verified by a positive pregnancy test
* Known hypersensitivity to the IMPs or any of their formulation ingredients
* Subject who is imprisoned or is lawfully kept in an Institution
* Employee or direct relative of an employee of the study site or the Sponsor
* Participation in an interventional clinical study with an IMP within the last 4 weeks before Screening
* Previous participation in this clinical study
* Planned extended stay outside the region which prevents compliance with the visit schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-10-19 (Estimated); Study Completion 2025-10-19 (Estimated)

PRIMARY OUTCOMES:
Presence of MDA (minimal disease activity) 12 months after baseline. | 12 months
  The MDA status comprises the assessment of different domains of PsA, consisting of the following individual components:
  * swollen and tender joint count
  * tender entheseal point count
  * skin involvement (PASI)patient self-assessment of pain (VAS)
  * global disease activity status
  * subject's self-assessment of functional ability using Stanford Health Assessment Questionnaire disability index, (HAQ-DI)
  MDA is defined as the presence of 5 of the following 7 criteria:
  1. tender joint count ≤1
  2. swollen joint count ≤1
  3. tender entheseal point count ≤1 (means: remission)
  4. PASI ≤1 OR body surface area (BSA) ≤3%
  5. patient pain VAS ≤15
  6. patient global activity VAS ≤20
  7. HAQ-DI ≤0.5

SECONDARY OUTCOMES:
Key secondary endpoint: PASDAS (Psoriatic Arthritis Disease Activity Score) | 12 months
  The PASDAS is a composite disease activity index (range 0-10) for psoriatic arthritis (PsA) incorporating seven domains: patient and physician global activity VAS scores, tender and swollen joint counts (arthritis), dactylitis, enthesitis (Leeds), health-related QoL (SF-36), and CRP level. PASDAS has demonstrated to have a better discriminate capacity in distinguishing high and low disease activity. The PASDAS is computed by the following equation: PASDAS = (((0, 18 ∗
  ∗√(PhGA) + 0.159 ∗ ∗√(PtGA) - 0.253 ∗ ∗√(SF36 -PCS) + 0.101 ∗ lognat(SJC66 + 1)) + 0.048 ∗ lognat(SJC68 +1)) + 0.23 ∗ lognat (Leeds enthesitis index + 1)) + 0.37 ∗lognat (tender dactylitis count + 1) + 0.102 ∗ lognat (CRP +1) + 2 ∗ 1.5.
Key secondary endpoint: DAPSA (Disease Activity in PSoriatic Arthritis) | 12 months
  The DAPSA score determines changes in the disease activity of subjects diagnosed with PsA. DAPSA is a composite score which is calculated from the sum of: number of tender joints (0-68), number of swollen joints (0-66, hips are not taken into account), CRP (mg/dl), subject's assessment of global status of disease activity using VAS (0-10) and patient's self-assessment of pain using VAS (0-10). A value of the composite score DAPSA 0-≤ 4 marks remission, 5-14 marks low, 15-28 moderate and >28 high disease activity
Key secondary endpoint: CPDAI (Composite Psoriatic Disease Activity Index) | 12 months
  The composite psoriatic disease activity index (CPDAI) assesses disease activity under five domains using well established and validated instruments of PsA disease documentation as proposed by GRAPPA. The domains and the respective instrument are as follows: joint disease (SJC/TJC, HAQ), skin involvement (PASI, DLQI), enthesitis (LEI, HAQ), dactylitis (dactylitis digit count, HAQ) and spinal involvement (BASDAI and ASQoL). Using the instruments and ranges of values, disease activity under each domain is graded as none (0) -mild (1) -moderate (2) and severe (3) giving a range attainable CPDAI scores of between 0 and 15. The CPDAI correlates well with patient and physician global disease activity assessments and is an effective tool that clearly distinguishes those who require a treatment change from those who do not.
Number of swollen and tender joints | 12 months
  An assessment of 66 joints for swelling and 68 joints for tenderness will be made (including the DIP joints of the hands and excluding hips for swelling).
Number of tender entheseal points: SPARCC (Spondyloarthritis Consortium of Canada) | 12 months
  The SPARCC enthesitis score is based on the counting of the presence or absence of tenderness on 16 entheseal sites (eight sites on each body side, respectively): lateral epicondyle, medial epicondyle, supraspinatus insertion into greater tuberosity of humerus, greater trochanter, quadriceps insertion into superior borders of patella, patellar ligament insertion into inferior pole of patella or tibial tubercle, Achilles tendon insertion into calcaneum, and plantar fascia insertion into calcaneum. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 16 sites, summarized in an overall score ranging from 0 to 16. A higher count represents a greater enthesitis burden
Number of tender entheseal Points: LEI (Leeds Enthesitis Index) | 12 months
  The LEI includes 3 entheseal sites on each body side, respectively: lateral epicondyles, medial condyles of the femur, and Achilles tendons. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 6 sites, for in an overall score ranging from 0 to 6. A higher count represents a greater enthesitis burden
Number of tender entheseal Points: MASES (Maastricht Ankylosing Spondylitis Enthesitis Score) | 12 months
  The MASES includes 6 entheseal sites on each body side (first costochondral joints, seventh costochondral joints, posterior superior iliac spines, anterior superior iliac spines, iliac crests, proximal insertion of Achilles tendons) and in addition the fifth lumbar spinous process. Tenderness on examination is recorded as either present (1) or absent (0) for each of the 13 sites, for an overall score ranging from 0 to 13. A higher count represents a greater enthesitis burden
Dactylitis counts | 12 months
  The presence of dactylitis will be assessed by counting the fingers/toes with dactylitis.
Activity of psoriasis: PASI (Psoriasis Area and Severity Index) | 12 months
  PASI combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 (no disease) to 72 (maximal disease).
Activity of psoriasis: BSA (body surface area) | 12 months
  For the BSA assessment of psoriatic skin involvement the size of the subject's hand is used as a scale to estimate the size of the skin surface covered by psoriasis. The subject's palm covers roughly 1% of body's surface area. An involved area of <3% of the skin is considered as mild, of 3 10% as moderate, and >10% as severe psoriasis
Activity of axial Involvement: BASDAI (Disease Activity of Ankylosing Spondylitis) | 12 months
  The BASDAI consists of a one through 10 scale (one being no problem and 10 being the worst problem) which is used to answer 6 questions pertaining to the 5 major symptoms of AS: Fatigue, Spinal pain, Joint pain / swelling, areas of localized tenderness (also called enthesitis, or inflammation of tendons and ligaments), morning stiffness duration, morning stiffness severity.
  To give each symptom equal weighting, the mean (average) of the two scores relating to morning stiffness is taken. The resulting 0 to 50 score is divided by 5 to give a final 0 - 10 BASDAI score. Scores of 4 or greater suggest suboptimal control of disease, and patients with scores of 4 or greater are usually good candidates for either a change in their medical therapy or for enrollment in clinical trials evaluating new drug therapies directed at Ankylosing Spondylitis
Quality of life and health/disability: PsAID-12 (Psoriatic Arthritis Impact of Disease) | 12 months
  The PsAID-12 is a score based on a subject's self-assessment questionnaire and used to measure the impact of psoriatic arthritis on a person's life. The questionnaire comprises 12 numeric rating scale questions covering the following topics: pain, fatigue, skin problems, work/leisure activities, functional capacity, discomfort, sleep disturbance, coping with PsA, anxiety and fear and uncertainty, embarrassment and/or shame, social participation, depression. Each question receives a score from 0 to 10. For evaluation these are weighted by factors and then summarized. The range of the final PsAID-score will be 0-10 where higher figures indicate worse status.
Quality of life and health/disability: HAQ-DI (Stanford Health Assessment Questionnaire Disability Index) | 12 months
  The Stanford Health Assessment Questionnaire is based on a subject's self-assessment questionnaire for persons diagnosed with PsA. The HAQ-DI assesses a patient's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in eight categories of functioning which represent a comprehensive set of functional activities - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The stem of each item asks for the past week "Are you able to …" perform a particular task. The patient's responses are made on a scale from zero (no disability) to three (completely disabled). Each category contains at least two specific component questions.
Quality of life and health/disability: DLQI (Dermatology Life Quality Index) | 12 months
  The DLQI is a score based on a subject's self-assessment questionnaire and used to measure the impact of the skin disease (psoriasis) on the quality of life of an affected person. The questionnaire contains 10 questions covering the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question refers to the impact of the skin disease on the patient's life over the previous week. Each question receives a score from 0 to 3. These are summarized to a final score with a possible range from 0 (meaning no impact on quality of life) to 30 (meaning maximum impact on quality of life).
Quality of life and health/disability: ASQoL (Ankylosing Spondylitis Quality of Life) | 12 months
  The ASQoL is a scale based on a subject's self-assessment questionnaire to measure the impact of ankylosing spondylitis (AS) on the quality of life of a diseased person with emphasis on the ability of the person to fulfill his or her needs. It consists of 18 items requesting a yes or no response to questions related to the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. The score range is 0-18. High scores indicate worse quality of life.
Quality of life and health/Disability: SF-36 (Short Form Health) | 12 months
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized for routine monitoring and assessment of care outcomes in adult patients. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. The eight sections are: vitality, physical functioning, bodily pains, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Pain (VAS) | 12 months
  The subject will be asked to place a vertical line on a 100-mm scale on which the left-hand boundary represents "no pain," and the right-hand boundary represents "pain as severe as can be imagined." The distance from the mark to the left-hand boundary will be recorded
Proportion of patients with loss of MDA within 12 months after baseline | 12 months
Proportion of patients with loss of MDA within 24 months after baseline | 24 months
Time to loss of MDA | 12 months
Time needed to restore MDA after readjustment of the DMARD therapy in subjects who lost MDA within the intervention period | 12 months
  Time [days/weeks/month] to restore after lost MDA
Biomarker levels | 24 months
  Serum cytokines, and molecular characterization of peripheral blood cells (e.g. IL-8 (CXCL8), Calprotectin (S100A9/S100A9). IL-22, lipocalin-2 (NGAL), beta defensin 2 [11], ILC, PBMC)
Intervention-related events within the observation period of 24 months after baseline | 24 months
  Observed symptoms (AE) related to reduction (intervention) such as symptoms suspicious of worsening disease activity (flare)
AE (Adverse Event) | 12 months
  Adverse Event
AR (Adverse Reaction) | 12 months
  Adverse Reaction
SAE (Serious Adverse Event) | 12 months
  Serious Adverse Event
SAR (Serious Adverse Reaction) | 12 months
  Serious Adverse Reaction
SUSAR (Suspected Unexpected Serious Adverse Reaction) | 12 months
  Suspected Unexpected Serious Adverse Reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
After all data of the trial were published by the study group, the data might be provided to interested scientists on request (e.g. for meta-analyses, health related registers or other scientific questions) in an anonymized way, if the members of the study group agree.